CLINICAL TRIAL: NCT02314429
Title: Phase I Trial Evaluating the Safety of a Lactate Releasing Vaginal Ring for the Prophylaxis of Bacterial Vaginosis
Brief Title: Trial Evaluating the Safety of a Lactate Releasing Vaginal Ring for the Prophylaxis of Bacterial Vaginosis
Acronym: LACRING01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Organization: University Hospital, Ghent (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: EC 2013/088; 2013-001120-19 (EudraCT Number)
Record Dates: First submitted 2014-12-02; First posted 2014-12-11 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Vaginosis, Bacterial
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaginal Ring (Experimental): A vaginal ring that slowly releases lactic acid (racemic mixture) into the vaginal environment, will be inserted in healthy volunteering women and left in place for 7 days.
  Interventions: Device: Vaginal ring releasing lactic acid (racemic mixture)

INTERVENTIONS:
Device: Vaginal ring releasing lactic acid (racemic mixture)

SUMMARY:
In this first-in-human volunteer phase I clinical trial, a vaginal ring that slowly releases lactic acid (racemic mixture) into the vaginal environment, will be inserted in healthy volunteering women and left in place for 7 days. The primary objective of this phase I study is to assess the safety and the tolerability of this new intravaginal delivery system.

The eventual goal of this and related studies is to develop a vaginal ring that reduces recurrences in women suffering from bacterial vaginosis, which is the commonest form of vaginal infection.

ELIGIBILITY:
Inclusion Criteria:

* Good general physical and mental health
* Presence of normal (lactobacilli-dominated) vaginal microbiota
* Prepared to take oral contraception during the study

Exclusion Criteria:

* Pregnancy
* Lactation
* Systemic disease
* Menopause
* Recent use of antibiotics (<1 week before entering the study)
* Recent use of intravaginal products or devices (<1 week before enrolment)
* Presence of vaginal infection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Absence/presence of visible cervicovaginal inflammation/irritation by colposcopy | 1 hour after insertion
Absence/presence of visible cervicovaginal inflammation/irritation by colposcopy | 2 hours after insertion
Absence/presence of visible cervicovaginal inflammation/irritation by colposcopy | 4 hours after insertion
Absence/presence of visible cervicovaginal inflammation/irritation by colposcopy | 8 hours after insertion
Absence/presence of visible cervicovaginal inflammation/irritation by colposcopy | 24 hours after insertion
Absence/presence of visible cervicovaginal inflammation/irritation by colposcopy | 7 days after insertion

SECONDARY OUTCOMES:
Assessment of vaginal pH | each 30 minutes for 4 hours after insertion, and then each 60 minutes for the next 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hans Verstraelen, Prof. dr., Principal Investigator — University & University Hospital Ghent
Locations (1):
- Department of Obstetrics & Gynaecology, Ghent University Hospital P4, Ghent, Belgium

REFERENCES:
- [Derived] Verstraelen H, Vervaet C, Remon JP. Rationale and Safety Assessment of a Novel Intravaginal Drug-Delivery System with Sustained DL-Lactic Acid Release, Intended for Long-Term Protection of the Vaginal Microbiome. PLoS One. 2016 Apr 19;11(4):e0153441. doi: 10.1371/journal.pone.0153441. eCollection 2016. PMID 27093291